CLINICAL TRIAL: NCT06749769
Title: Investigation of the Effectiveness of Simulation-Based Learning Experience in Strengthening Stoma Care Education on Patients With Stoma
Brief Title: Simulation-Based Learning Experience in Strengthening Stoma Care Education
Acronym: SIMESEP
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to changes in the clinical research team. The surgeon responsible for performing the study-related procedures has left the study hospital. The research team is currently seeking an appropriately qualified investigator to resume the study.
Sponsor: Nuran Ayşen Pamir Aksoy (Other)
Responsible Party: Sponsor-Investigator, Nuran Ayşen Pamir Aksoy, Assist. Prof., Acibadem University
Organization: Acibadem University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-17/648
Record Dates: First submitted 2024-12-16; First posted 2024-12-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Stoma
Keywords: stoma care; patient education; simulation; patient's learning experience; Strengthening patients

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients in the control group will receive routine verbal instructions and demonstration education about their stoma care.
- Study Group (Experimental): Participants in this group will receive a simulation-based stoma care education.
  Interventions: Behavioral: simulation-based education

INTERVENTIONS:
Behavioral: simulation-based education — Patients will learn how to care for their stomata on a stoma simulator
  Arms: Study Group

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of simulation-based learning experience in enhancing stoma care education on patients with stoma.

The main hypothesis it aims to test are:

H1: Simulation-based learning experience is effective in reducing stoma patients' concerns about performing stoma care.

H2: Simulation-based learning experience is effective in increasing stoma patients' stoma care skills.

H3: Simulation-based learning experience is effective in increasing stoma patients' perceived self-efficacy regarding stoma care.

Researchers will compare the control and study group to see if the simulation-based learning enhances the patients learning experience.

Participants will be asked to;

* Answer the questions (demographic data form and anxiety scale)
* Receive education regarding stoma care (verbal and demonstration)
* Practice stoma care on their own

ELIGIBILITY:
Inclusion criteria

1. Age 18 and above
2. First time having a stoma and having an intestinal stoma,
3. Communicable, open to cooperation,
4. Able to speak and understand Turkish,
5. Individuals who are willing to participate in the research and willing to be interviewed will be included in the research.

Exclusion Criteria

1. Patients who develop surgical complications in their stoma.
2. Patients who are unable to perform stoma care due to any complication
3. Having previously received stoma care training or participated in its implementation for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Stoma Care Skills Rubric | Post-operative 3rd day
  It consists of 23 items that include stoma care process steps. The learner's competence for each process step is scored between 0-2 (0- Insufficient 1- Partially sufficient 2- Sufficient). A minimum of 0 and a maximum of 46 points can be obtained. The total score shows the competence of stoma care skills.
Generalized Perceived Self-Efficacy Scale | at the time of enrollement, and Post-operative 3rd day
  It consists of 10 items, and each item of the scale is scored between 1 and 4. These are listed as not true (1), somewhat true (2), more true (3), and completely true (4). Minimum of 10 and a maximum of 40 points can be obtained. The higher the score, the higher the individual's perceived self-efficacy.

SECONDARY OUTCOMES:
State Anxiety Level | at the time of enrollement, and post-operative 3rd day
  In the study, the state anxiety scale will be used to determine the anxiety levels of the patients during the application. The State Anxiety Scale (SAS) provides information about what the individual feels at that moment. The State Anxiety Scale is a Likert-type scale consisting of 20 items, rated between 1 (not at all) and 4 (completely).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Acibadem Altunizade Hospital, Istanbul, Other
  - Acibadem Atakent Hospital, Istanbul, Other

IPD SHARING:
Plan to Share IPD: Undecided